CLINICAL TRIAL: NCT01316744
Title: A Randomized Double-Blind Controlled Trial of Ketamine Versus Placebo in Conjunction With Best Pain Management in Neuropathic Pain in Cancer Patients
Brief Title: Ketamine Hydrochloride and Best Pain Management in Treating Cancer Patients With Neuropathic Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000696704; CRUK-KPS-2008-01; EU-21012; EUDRACT-2007-002080-27; ISRCTN-49116945
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-03

CONDITIONS: Cancer
Keywords: long-term effects secondary to cancer therapy in adults; anxiety disorder; depression; pain; unspecified adult solid tumor, protocol specific; neuropathy; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression; Pain; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis; Myeloproliferative Disorders | interventions — Ketamine; Pharmacogenomic Testing

INTERVENTIONS:
Drug: ketamine hydrochloride
Other: pharmacogenomic studies
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Ketamine hydrochloride may lessen neuropathic pain in patients with cancer. It is not yet known whether ketamine hydrochloride given together with the best pain management is more effective than a placebo given together with the best pain management in treating neuropathic pain in patients with cancer.

PURPOSE: This randomized phase III trial is studying ketamine hydrochloride given together with the best pain management to see how well it works compared with giving a placebo together with the best pain management in treating cancer patients with neuropathic pain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether ketamine hydrochloride given in addition to best standard pain management improves malignant neuropathic pain compared to best standard pain management alone in patients with cancer.

Secondary

* To compare initial treatment benefit (at day 4 of assessment period of 16 days) using the sensory component of the McGill Short-Form Questionnaire.
* To compare difference in overall pain between the study arms based on the pain-intensity visual-analogue score (VAS).
* To compare difference in neuropathic pain between the study arms based on the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale.
* To assess worst pain score (index neuropathic site) between the two arms.
* To compare patient distress between the two arms based on NCCN Distress Thermometer.
* To assess the side effects and tolerability of trial drug.
* To assess the effect of intervention on quality of life scores (based on Euroqol thermometer), anxiety and depression (based on HADS), and opioid requirements.

OUTLINE: This is a multicenter study.

* Stage 1 (Run-in Period): Opioid doses are optimized, under a defined schedule, for up to a maximum of 10 days to ensure that all patients are on an optimized and stable regimen* prior to randomization. Following the run-in-period, patients undergo reassessment. Patients who have improved pain scores (i.e., < 4/10 on the visual-analogue score in the past 24 hours or < 5 McGill Sensory Scale Score) are taken off the study. Patients whose scores have not improved continue on to Stage 2 of the study.

NOTE: *Stable regimen is defined as the same dose of controlled release and no more variation than 2 breakthrough opioid doses over the normal for that patient for a period of 48 hours.

* Stage 2 (Titration Period): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral ketamine hydrochloride 4 times a day. Doses are titrated until when analgesia is achieved or individual side effects appear, for up to 14 days.
  * Arm II: Patients receive an oral placebo 4 times a day. Doses are titrated until when analgesia is achieved or individual side effects appear, for up to 14 days.
* Stage 3 (Assessment Period): Patients receive the trial medication (i.e., ketamine hydrochloride or placebo) at the fixed optimum dose (reached during the titration period) for 16 days.

Patients are allowed to receive breakthrough opioids at any time during the study.

Patients complete quality-of-life and pain-assessment questionnaires periodically. Some patients may undergo blood sample collection periodically for pharmacogenomics studies at a later date.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer
* Index neuropathic pain ≥ 4 on 0-10 (as defined by Leeds Assessment of Neuropathic Symptoms and Signs) that is related to underlying malignancy or resulting from treatment received for this malignancy
* McGill Sensory Scale Score > 5
* Received a trial of an adjuvant analgesic (gabapentin or amitriptyline or both)

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 2 months
* Fertile patients must use effective contraception
* Able to comply with study procedures
* Diastolic blood pressure ≤ 100 mm Hg at screening
* No seizures in past 2 years
* Not actively hallucinating
* No cerebrovascular disease (strokes)
* No psychotic disorders or cognitive impairment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior and no concurrent chemotherapy or radiotherapy that is likely to affect neuropathic pain
* No change in tumoricidal treatment during the period of the study that is likely to alter pain during the course of the study
* No concurrent class I antiarrhythmic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure

SECONDARY OUTCOMES:
Initial treatment benefit (at day 4 of assessment period of 16 days) using the sensory component of the McGill Short-Form Questionnaire
Difference in overall pain between the study arms based on the visual-analogue score
Difference in neuropathic pain between the study arms based on the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale
Worst pain score (index neuropathic site) in the previous 24 hours (between the two arms) at study baseline and then during study assessment period
Patient distress between the two arms based on NCCN Distress Thermometer
Side effects and tolerability of trial drug
Effect of the intervention on quality-of-life scores (based on Euroqol thermometer), anxiety and depression (based on HAD scale), and opioid requirements

CONTACTS AND LOCATIONS:
Overall Officials: Marie T. Fallon, Principal Investigator — Edinburgh Cancer Centre at Western General Hospital; Barry J.A. Laird, MD, Principal Investigator — Edinburgh Cancer Centre at Western General Hospital
Locations (3):
- United Kingdom (3):
  - Royal Brompton Hospital, London, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland